CLINICAL TRIAL: NCT05769036
Title: Randomized Study of Integrated Evaluation of Conventional Biventricular and Left Bundle Branch Pacing Therapy Effect on Left Ventricular Remodeling and Clinical Outcomes in Patients With Chronic Heart Failure With Reduced Ejection Fraction
Brief Title: Conventional Biventricular Versus Left Bundle Branch Pacing on Outcomes in Heart Failure Patients
Acronym: RECOVER-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Principal Investigator, Tariel A. Atabekov, Principal Investigator, Tomsk National Research Medical Center of the Russian Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECOVER-HF
Record Dates: First submitted 2023-02-20; First posted 2023-03-15 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Left Bundle-Branch Block; Ischemic Cardiomyopathy; Non-ischemic Dilated Cardiomyopathy; Left Ventricular Dysfunction; Left Ventricular Dyssynchrony; Left Ventricle Remodeling
Keywords: Cardiac Resynchronization Therapy; Biventricular Pacing; Left Bundle Branch Pacing; Speckle Tracking Echocardiography; Biomarker of Fibrosis and Remodeling
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block; Ventricular Dysfunction, Left; Ventricular Remodeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cardiac Resynchronization Therapy with Biventricular Pacing (Active Comparator): Patients in this group will be implanted with a cardioverter-defibrillator with a resynchronization function using the biventricular pacing
  Interventions: Device: Implantation of Cardioverter-defibrillator with a Resynchronization Function Using Biventricular Pacing
- Cardiac Resynchronization Therapy with Left Bundle Branch Pacing (Experimental): Patients in this group will be implanted with a cardioverter-defibrillator with a resynchronization function using the left bundle branch pacing
  Interventions: Device: Implantation of Cardioverter-defibrillator with a Resynchronization Function Using Left Bundle Branch Pacing

INTERVENTIONS:
Device: Implantation of Cardioverter-defibrillator with a Resynchronization Function Using Biventricular Pacing — The local anesthesia will be performed on the left/right subclavian area after prepping the skin. A horizontal incision will be performed. The cephalic and subclavian veins will be used to leads deliver. The active-fixation defibrillation lead will be placed to the apex/interventricular septum. The atrial active-fixation lead will be implanted to the right atrial appendage/interatrial septum. The implantation of the left ventricular pacing lead will be performed by cannulating one of the tributaries of the coronary sinus using delivery system. Leads will be fixated, connected with CRT-D device and placed in subcutaneous (subfascial prepectoral)/submuscular pocket. The pocket will be closed by separate stitches (2-4 suffice) using the resorbable braided suture. Cardioverter-defibrillator with a resynchronization function will be programmed for biventricular pacing.
  Arms: Cardiac Resynchronization Therapy with Biventricular Pacing
Device: Implantation of Cardioverter-defibrillator with a Resynchronization Function Using Left Bundle Branch Pacing — The local anesthesia will be performed on the left/right subclavian area after prepping the skin. A horizontal incision will be performed. The cephalic and subclavian veins will be used to leads deliver. The active-fixation defibrillation lead will be placed to the apex/interventricular septum. The atrial active-fixation lead will be implanted to the right atrial appendage/interatrial septum. The implantation to the left bundle branch will be performed by using special delivery system. Leads will be fixated, connected with CRT-D device and placed in subcutaneous (subfascial prepectoral)/submuscular pocket. The pocket will be closed by separate stitches (2-4 suffice) using the resorbable braided suture. Cardioverter-defibrillator with a resynchronization function will be programmed left bundle branch pacing.
  Arms: Cardiac Resynchronization Therapy with Left Bundle Branch Pacing

SUMMARY:
Heart failure (HF) is the most common nosology encountered in clinical practice. Its incidence and prevalence increase exponentially with increasing age and it is associated with increased mortality, more frequent hospitalization and decreased quality of life. An initial approach to the treatment of HF patients with reduced left ventricular (LV) systolic function and left bundle branch block (LBBB) was implantation of cardioresynchronization device using biventricular pacing. This has resulted in long-term clinical benefits such as improved quality of life, increased functional capacity, reduced HF hospitalizations and overall mortality. However, conventional cardiac resynchronization therapy (CRT) is effective in only 70% of patients. And the remaining 30% of patients are non-responders to conventional CRT. Subsequently, His bundle pacing (HBP) has been developed to achieve the same results. According to other studies HBP has showed greater improvement in hemodynamic parameters than with conventional biventricular CRT. But, nevertheless, there are significant clinical troubles with HBP. In this regard, in 2017, the left bundle branch pacing (LBBP) was developed, which demonstrated clinical advantages compared to biventricular CRT. This method has become an alternative to HBP due to the stimulation of LBB outside the blocking site, a stable pacing threshold and a narrow QRS duration. A series of case reports and observational studies have demonstrated the efficacy and safety of LBBP in patients with CRT indications. However, it is not enough data about CRT with LBBP effectiveness in LV remodeling, reducing mortality and complications. According to our hypothesis, CRT with LBBP compared with conventional biventricular CRT will significantly improve the clinical outcomes and reverse LV remodeling in patients with chronic HF with reduced LV ejection fraction and reduce the number of non-responders to conventional CRT.

DETAILED DESCRIPTION:
The heart failure (HF) is a rapidly growing public health issue with an estimated prevalence of more than 37.7 million individuals globally. In the developed world, this disease affects approximately 2.0% of the adult population. In the United States the total percentage of the population with HF is projected to rise from 2.4% in 2012 to 3.0% in 2030. In Russian Federation the prevalence of chronic HF (CHF) is 10.2%. The main cause of CHF is a coronary heart disease, which accounts for about 70.0%, and the remaining 30.0% are non-ischemic heart diseases. More than 2 decades of research has established the role of cardiac resynchronization therapy (CRT) in medically refractory, mild to severe systolic HF with abnormal QRS duration and morphology. The prolongation of QRS (120 ms or more) occurs in 14.0% to 47.0% of HF patients and the ventricular conduction disturbance, most commonly left bundle branch block (LBBB), is present in approximately one-third of HF, leading to mechanical dyssynchrony of ventricles. Prospective randomized studies of patients with both ischemic HF (IHF) and non-ischemic HF (NIHF) have shown that CRT translates into long-term clinical benefits, such as improved quality of life, increased functional capacity, reduction in hospitalization for HF, and overall mortality. These patients qualified as responders to CRT. However, CRT is effective in 70.0% of patients, and the remaining 30.0% do not respond to the device therapy. In fact, biventricular CRT leads to the fusion of two fronts of non-physiological excitation waves and leaves a significant residual dyssynchrony.

His bundle pacing (HBP) is possible alternative to biventricular CRT. During HBP there is a physiological electromechanical synchrony by facilitating conduction through the native His-Purkinje system. HBP promotes higher electrical ventricular resynchronization than biventricular CRT. Studies have shown that HBP, as well as conventional biventricular CRT, improves cardiac function, which leads to a decrease in the number of HF hospitalizations. The main unsolved problems that limit the use of HBP are the low amplitude of the intracardiac signal, high pacing thresholds and troubles associated with lead implantation in the area of the His bundle, which ultimately increases the risk of re-implantation.

In 2017, W. Huang et al. pioneered left bundle branch pacing (LBBP) and demonstrated that it provided clinical benefits in patients with HF and LBBB, aiming to pacing the proximal left bundle branch (LBB) along with LV myocardial capture. During selective pacing, only LBB is captured without the nearby myocardium, while with non-selective LBBP the septal myocardium is captured. LBBP with lead implanted slightly distal to the His bundle and screwed deep into the left ventricular (LV) septum is ideal for the LBB capture. LBBP has emerged as an alternative to HBP due to pacing of LBB outside the blocking site, a stable pacing threshold, and a narrow QRS in patients with bradycardia. In clinical cases of W. Huang et al. was demonstrated for the first time that LBBP could lead to complete correction of LBBB and improvement in cardiac function in patients with LBBB and HF. In another observational study, W. Zhang et al. showed that LBBP could be a new method of CRT. Subsequently, several case reports and observational studies have demonstrated the efficacy and safety of LBBP in patients with indications for CRT device implantation.

The above studies demonstrate that LBBP is clinically feasible in patients with HF and LBBB. However, there are still few data about CRT using LBBP in patients with HF and reduced LVEF. There are also few studies on direct comparison of changes in clinical, speckle tracking echocardiography and other laboratory and instrumental parameters between patients with conventional biventricular CRT and CRT using LBBP.

CRT induces reverse remodeling of the affected heart, improves LV systolic and diastolic function and left heart filling pressure. The measurement of fibrosis and remodeling biomarkers representing the pattern of active processes in HF be useful.

The relationship between changes in the biomarkers level and reverse remodeling process in patients with LBBP is currently poorly understood. And there are no publications regarding the correlation of the level of such biomarkers as MR-proANP, GDF-15, galectin-3, ST2, MR-proADM and PINP with clinical and instrumental indicators of patients with LBBP in the available literature. This creates all the prerequisites for studying the association of the above biomarkers with the reverse remodeling process in patients with CRT using LBBP.

ELIGIBILITY:
Inclusion criteria:

1. The patient is willing and able to comply with the protocol and has provided written informed consent;
2. Male or female patients aged 18 to 80 years;
3. Patients with ischemic or non-ischemic cardiomyopathy;
4. Symptomatic HF for at least 3 months prior to enrollment in the study;
5. New York Heart Association (NYHA) functional class HF ≥ II;
6. Patients with HF in sinus rhythm (SR) with LVEF ≤ 35% (measured in the last 6 weeks prior to enrollment), QRS duration ≥150 ms with LBBB morphology;
7. Patients with HF in SR with LVEF ≤ 35% (measured in the last 6 weeks prior to enrollment), QRS duration 130-149 ms with LBBB morphology;
8. Patients with HF in SR with LVEF ≤ 35% (measured in the last 6 weeks prior to enrollment), QRS duration ≥150 ms with non-LBBB morphology;
9. Patients with symptomatic persistent or permanent atrial fibrillation, HF with LVEF < 40% (measured in the last 6 weeks prior to enrollment) and an uncontrolled heart rate who are candidates for atrioventricular junction ablation (irrespective of QRS duration);
10. Patients with HF, LVEF < 40% (measured in the last 6 weeks prior to enrollment) and indications for continuous ventricular pacing due to bradycardia;
11. Patients who have received a conventional pacemaker or an implanted cardioverter-defibrillator and who subsequently develop symptomatic HF with LVEF < 40% (measured in the last 6 weeks prior to enrollment) despite optimal medical therapy, and who have a significant proportion of right ventricle pacing;
12. Optimal HF medical therapy.

Exclusion criteria:

1. Coronary artery (CA) bypass grafting, balloon dilatation or CA stenting within 3 months prior to enrollment;
2. Acute myocardial infarction within 3 months prior to enrollment;
3. Acute coronary syndrome;
4. Patients with planned cardiovascular intervention (CA bypass grafting, balloon dilatation or CA stenting);
5. Patients listed for heart transplant;
6. Patients with implanted cardiac assist device;
7. Acute myocarditis;
8. Infiltrative myocardial disease;
9. Hypertrophic cardiomyopathy;
10. Severe primary stenosis or regurgitation of the mitral, tricuspid and aortic valves;
11. Woman currently pregnant or breastfeeding or not using reliable contraceptive measures during fertility age;
12. Mental or physical inability to participate in the study;
13. Patients unable or unwilling to cooperate within the study protocol;
14. Patients with rheumatic heart disease;
15. Mechanic tricuspid valve patients;
16. Patients with any serious medical condition that could interfere with this study;
17. Enrollment in another investigational drug or device study;
18. Patients not available for follow-up;
19. Patients with severe chronic kidney disease (estimated glomerular filtration rate ˂ 30 ml/min/1.73 m2);
20. Life expectancy ≤ 12 months;
21. Participation in another telemonitoring concept.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality or worsening of heart failure requiring unplanned hospitalization (%) | 24 months
  Definition of all-cause mortality All deaths and all heart transplants due to the terminal heart failure. Heart transplanted patients will be dropped out and followed in respect of their vital status for the duration of the study.
  Definition of worsening of heart failure requiring unplanned hospitalization Patients requiring intra-venous medication for heart failure (including diuretics, vasodilators or inotropic agents) or a substantial increase in oral diuretic therapy for heart failure (i. e. an increase of Furosemide ≥ 40 mg or equivalent, or the addition of a thiazide to a loop diuretic) will be deemed to have worsening of heart failure. Further, rales and/or S3 sound, chest x-ray, worsening of dyspnoea, worsening of peripheral edema and increase of class NYHA will be assessed for determination of worsening of heart failure. Unplanned hospitalization is defined as any in-hospital stay over one date change, and not planned by the Investigator.

SECONDARY OUTCOMES:
All-cause Mortality (%) | 24 months
  As defined for primary endpoint: all deaths and all heart transplants because of terminal heart failure.
Cardiovascular Mortality (%) | 24 months
  All deaths due to cardiovascular reasons and all heart transplants because of terminal HF. Deaths due to worsening of HF, acute coronary syndrome, cerebrovascular accidents, or other cardiovascular events will qualify for this secondary endpoint.
Worsening of Heart Failure Requiring Unplanned Hospitalization (%) | 24 months
  As defined for the primary end-point: patients requiring intra-venous medication for HF (including diuretics, vasodilators, or inotropic agents) or a substantial increase in oral diuretic therapy for HF (i. e. an increase of Furosemide ≥ 40 mg or equivalent, or the addition of a thiazide to a loop diuretic) will be deemed to have worsening of HF. Further, rales and/or S3 sound, chest x-ray, worsening of dyspnoea, worsening of peripheral edema, and increase of class NYHA will be assessed for determination of worsening of HF.
  Unplanned hospitalization is defined as any in-hospital stay over one date change, and not planned by the Investigator.
  Reasons for worsening of HF may include AF, acute coronary syndrome and hypertension.
Unplanned Hospitalization due to Cardiovascular Reason (%) | 24 months
  Any in-hospital stay over one date change due to cardiovascular reason, which includes worsening of HF, acute coronary syndrome, cerebrovascular accidents, or other cardiovascular events, and not planned by the Investigator.
  In case the hospitalization is classified as planned by the Investigator, and the time interval between the decision to hospitalize and the hospitalization is less than 24 hours.
All-cause Hospitalization (%) | 24 months
  Any in-hospital stay over one date change.
Number of Delivered CRT-D Shocks (n) | 24 months
  An CRT-D shock is an electrical treatment consisting of a high voltage capacitor discharge delivered upon detection of VT/VF episode. All ICD shocks will be collected and classified by the Investigator as successful or non successful in respect to the termination of the tachyarrhythmia.
Time to First CRT-D Shock (days) | 24 months
  It is the time interval between the end of the 12 weeks blanking after baseline and the first appropriate CRT-D shock in case of ventricular tachycardia or ventricular fibrillation.
Number of Delivered CRT-D ATPs (n) | 24 months
  An CRT-D antitachycardia pacing therapy (ATP) is an electrical treatment consisting of timed stimuli delivered upon detection of ventricular tachycardia/ventricular fibrillation (VT/VF) episode. All CRT-D ATPs will be collected and classified by the Investigator as successful or non successful in respect to the termination of the tachyarrhythmia.
Time to First CRT-D ATP (days) | 24 months
  It is the time interval between the end of the 12 weeks blanking after baseline and the first ATP therapy.
Number of Device Detected VT/VF Episodes (n) | 24 months
  It is any ventricular tachyarrhythmia which fulfils the programmed detection criteria of the device in order to be classified as tachyarrhythmic ventricular episode. Device detected episodes will be classified by the Investigator as appropriately detected in presence of real tachyarrhythmia, or inappropriately detected in case of other reasons (oversensing, noise, fast ventricular rate due to supraventricular tachycardia).
Left Ventricular Function (LVEF, %) | 24 months
  The measurement of the left ventricular ejection fraction performed by echocardiography using the modified Simpson's rule.
Exercise Tolerance (m) | 24 months
  It is the measurement of the maximal distance that the patient is able to walk within 6 minutes.
Life Quality (MLWHFQ score) | 24 months
  The life quality is the patient's ability to enjoy normal life activities. For patients suffering from HF, improvement of quality of life is one of the most important goals of new treatments, sometimes as important as improved survival. Some medical treatments can seriously impair quality of life without providing appreciable benefit, while others greatly enhance it. To evaluate the effect of cardiac resynchronization therapy with left bundle branch pacing on the quality of life of patients, general and heart failure-related quality of life questionnaires, both filled in by each individual patient, will be used.
  The Minnesota Living with Heart Failure Questionnaire (MLWHFQ, scale from 0 to 5) will be used.
Life Quality (EuroQoL EQ-5D score) | 24 months
  The life quality is the patient's ability to enjoy normal life activities. For patients suffering from HF, improvement of quality of life is one of the most important goals of new treatments, sometimes as important as improved survival. Some medical treatments can seriously impair quality of life without providing appreciable benefit, while others greatly enhance it. To evaluate the effect of cardiac resynchronization therapy with left bundle branch pacing on the quality of life of patients, general and heart failure-related quality of life questionnaires, both filled in by each individual patient, will be used.
  The European Quality of Life Questionnaire (EuroQoL EQ-5D, scale from 0 to 100) will be used.

OTHER OUTCOMES:
Echocardiography Left Ventricular Volume Improvement (%) | 24 months
  Echocardiographic measurements will be done at baseline, 6, 12, 18 and 24 month follow-up, to evaluate effect of CRT-D implantation on left ventricle (LV) volume. Improvements due to reverse remodelling of the heart will be evaluated by measuring left ventricular end-systolic volume (LVESV), which is supposed to decrease at follow-up. Further, LV volume improvment will be calculated using formula: ((A-B)/A) x 100% (A-baseline LVESV; B-follow-up LVESV).
Echocardiography Left Ventricular Ejection Fraction Improvement (%) | 24 months
  chocardiographic measurements will be done at baseline, 6, 12, 18 and 24 month follow-up, to evaluate effect of CRT-D implantation on left ventricle (LV) contractility function. Improvements due to reverse remodelling of the heart will be evaluated by measuring left ventricular ejection fraction (LVEF), which is supposed to increase at follow-up. Further, LV contractility function improvment will be calculated using formula: ((A-B)/A) x 100% (A-baseline LVEF; B-follow-up LVEF).
NYHA Class | 24 months
  The NYHA functional classification provides a simple way of classifying the extent of HF. It is based on questions, related to the usual daily activities and symptoms posed to the patients, and it will be determined at enrollment, baseline and at each FU visit. In ablated patients an improvement of NYHA class is expected, the analysis of which will help to assess the efficacy of ablation therapy.
Rate of Drug Support Requirements (%) | 24 months
  Beta-blockers, angiotensin-converting enzyme inhibitors, angiotensin II receptor antagonists, aldosterone antagonists, diuretics, and sodium-glucose transporter type 2 inhibitors, antiarrhythmics and diuretics are drugs commonly taken by patients suffering from HF. Those drugs may have the potential to induce AEs. In patients with left bundle branch pacing (LBBP) CRT-D a reduction in drug consumption is expected, with a consequent reduction of side effects. The evaluation of the drug regimen will help to assess the effectiveness of LBBP.

CONTACTS AND LOCATIONS:
Overall Officials: Tariel A Atabekov, Ph.D., Principal Investigator — Cardiology Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences; Roman E Batalov, M.D., Study Director — Cardiology Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences
Locations (1):
- Cardiology Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences, Tomsk, Russia